CLINICAL TRIAL: NCT06215261
Title: An Evaluation of the Safety and Efficacy of Methylone for the Treatment of PTSD IMPACT-2 (Investigation of Methylone for Post-Traumatic Stress Disorder [PTSD])
Brief Title: An Evaluation of the Safety and Efficacy of Methylone for the Treatment of PTSD
Acronym: IMPACT-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Transcend Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TSND201-PTSD-202
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Methylone; IMPACT-2; PTSD; Neuroplastogen; TSND-201
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — methylone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TSND-201 Low Dose (Experimental): Part B only
  Interventions: Drug: Methylone
- TSND-201 Mid Dose (Experimental): Part B only
  Interventions: Drug: Methylone
- TSND-201 High Dose (Experimental): Part B only
  Interventions: Drug: Methylone

INTERVENTIONS:
Drug: Methylone — Methylone capsules, given orally, once a week for 3 weeks (Part A) or 4 weeks (Part B)

SUMMARY:
This study is evaluating the safety and efficacy of methylone in adults with PTSD. The study is conducted in two parts.

* Part A is open-label and will enroll up to 15 participants with PTSD
* Part B is randomized (1:1:1), single-blind and will enroll up to 45 participants with PTSD

Eligible participants will enter a 3-week Treatment Period (Part A) or 4-week Treatment Period (Part B) where they will receive methylone once weekly. Following the Treatment Period, participants will enter a 6-week Follow-up Period (Part A) or 8-week Follow-up Period (Part B).

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-5 criteria for severe PTSD diagnosis, with a symptom duration of at least 6 months.
* Tried at least one treatment for PTSD (either psychotherapy or pharmacological treatment).
* Proficient in reading and writing in local language sufficient to complete questionnaires.
* Free from any other clinically significant illness or disease.

Exclusion Criteria:

* Primary diagnosis of any other DSM-5 disorder.
* Body mass index (BMI) <18kg/m2 or ≥40 kg/m2.
* Smokes an average of >10 cigarettes and/or e-cigarettes per day.
* Uncontrolled hypertension at Screening.
* Use of prohibited concomitant medications or therapies.
* Current or previous history of clinically significant cardiovascular/cerebrovascular conditions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Clinician-Administered PTSD Scale for the DSM-5 (CAPS-5) total severity score | 9 weeks (Part A) / 12 weeks (Part B)
  The CAPS-5 is a structured interview designed to assess PTSD symptom severity. The total severity score ranges from 0 to 80, with a higher score indicating more severe symptoms.

SECONDARY OUTCOMES:
Change from Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) total score | 9 weeks (Part A) / 12 weeks (Part B)
  The MADRS is a 10-item, clinician-rated scale designed to assess severity of depression. The total score ranges from 0 to 60, with a higher score indicating more severe depression.
Change from Baseline in PTSD Checklist for DSM-5 (PCL-5) | 9 weeks (Part A) / 12 weeks (Part B)
  The PCL-5 is a 20-item, patient-rated scale designed to measure severity of PTSD symptoms. The total score ranges from 0 to 80, with a higher score indicating more severe PTSD symptoms.
Change from Baseline in Sheehan Disability Scale (SDS) | 9 weeks (Part A) / 12 weeks (Part B)
  The SDS is a 3-item, patient-rated scale designed to measure disability and impairment across three domains: work/school, social life, and family life/home responsibilities. Each domain is scored from 0 to 10, with higher scores representing greater disability. Total scores range from 0 to 30.
Incidence of treatment-emergent adverse events (TEAEs) | 9 weeks (Part A) / 12 weeks (Part B)
  Types and rates of adverse events

CONTACTS AND LOCATIONS:
Locations (12):
- United States (8):
  - Segal Trials, Lauderhill, Florida
  - Accel Research, Maitland, Florida
  - CNS Healthcare, Orlando, Florida
  - Uptown Clinical Research, Chicago, Illinois
  - Sunstone Medical, Rockville, Maryland
  - Redbird Research LLC, Las Vegas, Nevada
  - Numinus, Draper, Utah
  - Seattle NTC, Bellevue, Washington
- Australia (3):
  - Swinburne University of Technology, Hawthorn, Victoria
  - Ramsay Clinic Albert Road, Melbourne, Victoria
  - Monarch Mental Health Group, Melbourne, Victoria
- Clerkenwell Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No